CLINICAL TRIAL: NCT02911181
Title: Quality Project Malnutrition Intensive Care
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Matty Koopmans, MSc, Frisius Medisch Centrum
Other Study IDs: nWMO 077
Record Dates: First submitted 2016-03-07; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Malnutrition
Keywords: BIVA measurement; SNAQ score
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: BIVA measurement

SUMMARY:
Observational study to investigate nutrition state in all admitted patients in ICU. Measurement by BIVA and SNAQ score.

DETAILED DESCRIPTION:
Malnutrition is a great problem in healthcare, its related to mortality, infections and length of stay. Observational study to investigate nutrition state in all admitted patients in ICU. Measurement by BIVA and SNAQ score.

All patients were asked for their nutrition state by SNAQ and the BIVA measurement is done by a trained doctor.

ELIGIBILITY:
Inclusion Criteria:

* admission ICU

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in the ICU between feb 2016 and may 2016
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
malnutrition | day 1 in Intensive Care
  percentage of patients with malnutrition at admission on the ICU

SECONDARY OUTCOMES:
malnutrition in elective and acute patients | day 1 in Intensive Care
  Is there a difference in malnutrition between elective patients and acute patients

CONTACTS AND LOCATIONS:
Overall Officials: Matty Koopmans, MSc, Principal Investigator — Intensive Care
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buter H, Veenstra JA, Koopmans M, Boerma CE. Phase angle is related to outcome after ICU admission; an observational study. Clin Nutr ESPEN. 2018 Feb;23:61-66. doi: 10.1016/j.clnesp.2017.12.008. Epub 2017 Dec 20. PMID 29460815